CLINICAL TRIAL: NCT04988022
Title: Defining Reversal of Keloid Lesions by Th2 Targeting With Dupilumab Treatment
Brief Title: Dupilumab in the Treatment of Keloids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Emma Guttman, Professor and Chair, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 20-3159
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dupilumab (Experimental): dupilumab 600mg loading dose at Baseline (given as two 300 mg injections) followed by one 300mg weekly subcutaneous injection through Week 52.
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): matching placebo loading dose at Baseline (given as two injections) followed by one weekly subcutaneous injection through Week 24. Starting at Week 24, dupilumab 600mg loading dose (given as two 300 mg injections) followed by one 300mg weekly subcutaneous injection through Week 52.
  Interventions: Drug: Dupilumab; Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — 300 mg prefilled syringe
  Other Names: Dupixent
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This study is a prospective, randomized, double blind, placebo-controlled clinical trial.

The study will include a total of 44 subjects with clinically measurable keloid lesions. At least 50% of subjects (at least 22 out of the 44 subjects) will also have documented diagnosis of concomitant type 2 atopic/allergic) inflammatory diseases. In Phase I, subjects will be randomized (3:1) to either receive weekly dupilumab or placebo for 24 weeks. At Week 24, both groups will enter Phase II of the study in which all subjects will receive weekly doses of dupilumab up to Week 52. The treatment period will conclude at Week 52.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double blind, placebo-controlled clinical trial.

The study will include a total of 44 subjects with clinically measurable keloid lesions. At least 50% of subjects (at least 22 out of the 44 subjects) will also have documented diagnosis of concomitant type 2 atopic/allergic) inflammatory diseases. In Phase I, subjects will be randomized (3:1) to either receive weekly dupilumab or placebo for 24 weeks. At Week 24, both groups will enter Phase II of the study in which all subjects will receive weekly doses of dupilumab up to Week 52. The treatment period will conclude at Week 52.

After providing consent, subjects will be assessed for study eligibility during the screening period (within 28 days of Baseline), which includes a review of the subject's past and current medical conditions as well as a family history of keloids, atopic dermatitis (AD), asthma and other atopic diseases, detailed review of past and current medications, review of past topical and systemic treatments/therapies and invasive treatments (including surgery, radiation, and cryotherapy) for keloids, limited physical examination, clinical assessments (number, location and measurements via tonometer and calipers). Measurements of keloid lesions will be standardized and performed using Verneir Calipers. These are accurate to the nearest 0.01mm in their measurement of all dimensions. Keloid distensibility (hardness) will be measured using a tonometer, a tool that has been adapted for use in systemic sclerosis and can give insight into softening of lesions.

Subjects who meet inclusion criteria for eligibility will undergo Baseline assessments at Week 0, including clinical assessments (number, location and measurements via tonometer and calipers), review of concomitant medications, standardized clinical photography, questionnaires (a Dermatology Life Quality Index (DLQI), and a Keloid-Quality of Life Index (K-QLI) questionnaire), and additional skin assessments if he/she concurrently has atopic dermatitis (EASI, IGA, BSA and SCORAD will be used to evaluate existing atopic dermatitis). Blood samples and skin biopsies will be collected for mechanistic studies (described below) at various timepoints for RNA, DNA and protein analyses, as well as for analyses of IgE and serum CRP. Two 4.5 mm biopsies will be performed at Baseline: one from a keloid lesion and one from an adjacent non-lesional area. Non-lesional biopsies will mimic nascent trauma (e.g. surgery, or other inflammatory processes) and evaluate the effectiveness of dupilumab in preventing new keloid lesion formation.

Subjects will return for visits at weeks 4, 8, 16, 24, 28, 36, 48, and 52 following study treatment initiation for repeat clinical assessments (number, location, and measurements via tonometer and calipers), medication reviews, blood and biopsy collection, surveys, and monitoring for adverse events. At week 24 a second lesional biopsy will be performed (from the same keloid area biopsy at baseline, but away from the previous biopsy scar), and at week 48 both a lesional (again from the same keloid, but away from prior biopsies) and a non-lesional biopsy will be performed. Bloods will be done at baseline, week 4, week 16, week 24, week 48. The biopsy sites as well as other lesional areas will be monitored at each subsequent visit by clinical assessment (number, location and measurements via tonometer and calipers) and standardized clinical photography.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥ 18 years of age at the time of signing the informed consent document.
* Subject is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures.
* Subject is able to adhere to the study visit schedule and other protocol requirements.
* Subject has at least two clinically measurable keloid lesions on the trunk and/or extremities, that failed prior minimally invasive treatments for keloids including topicals and intralesional steroid injections. However, at least one keloid should not have been treated with surgery, cryotherapy, radiation, or any other procedure that leads to a deformity that interferes with proper clinical assessments.
* At least 50% of the subjects: subject has documented diagnosis of concomitant type 2 (atopic/allergic) (e.g., active AD, asthma, chronic rhinosinusitis with nasal polyposis, food allergy confirmed by skin prick test or food allergen specific IgE, seasonal allergies, other confirmed allergies).
* Subject is judged to be in otherwise good overall health as judged by the investigator, based on medical history, physical examination, and laboratory testing. (NOTE: The definition of good health means a subject does not have uncontrolled significant co-morbid conditions).
* Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective contraceptive methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy.

OR

Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

The female subject's chosen form of contraception must be effective by the time the female subject is randomized into the study (for example, hormonal contraception should be initiated at least 28 days before randomization).

Exclusion Criteria:

* Subject has a persistent or recurring bacterial infection requiring systemic antibiotics, or clinically significant viral or fungal or helminth parasitic infections, within 2 weeks of the Screening Visit. Any treatment of such infections must have been completed at least 2 weeks prior to the Screening Visit and no new/recurrent infections should have occurred prior to the Baseline Visit.
* Subject with current or history of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (i.e. Common Variable Immunodeficiency [CVID]), hepatitis B or C, or active or untreated latent tuberculosis.
* Subject has clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other major uncontrolled diseases that will affect the health of the subject during the study, or interfere with the interpretation of study results.
* Subject has a suspected or active lymphoproliferative disorder or malignancy; OR a history of malignancy within 5 years before the Baseline assessment, except for completely treated in situ non-melanoma skin and cervical cancers without evidence of metastasis.
* Subject was treated previously with dupilumab.
* Subject has received a live attenuated vaccine ≤ 30 days prior to study initiation.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Severe, untreated asthma or a history of life-threatening asthma exacerbations while on appropriate regimen of anti-asthmatic medications.
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus, or ultraviolet (UV) phototherapy with or without Psoralen Ultraviolet A (PUVA) therapy within 4 weeks prior to trial initiation.
* Use of an oral JAK inhibitor (tofacitinib, ruxolitinib) within 12 weeks prior to the Baseline visit.
* Subject has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus on any keloid lesions within 1 week prior to the Baseline visit. These will be allowed during the study on areas of atopic dermatitis (if applicable) but not on any keloid lesions.
* Female subject who is pregnant or breast feeding
* Subject currently uses or plans to use anti-retroviral therapy at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in dimensions of keloid lesions at 24 weeks | baseline and 24 weeks
  Change from baseline in dimensions of keloid lesions (length, width, and depth in cm) at 24 weeks of treatment with dupilumab performed using Verneir Calipers.

SECONDARY OUTCOMES:
Change from baseline in dimensions of keloid lesions at weeks 4, 16, 24, 48, and 52 of treatment with dupilumab | baseline and weeks 4, 16, 24, 48, and 52
  Change from baseline in dimensions of keloid lesions (length, width, and depth in cm) at weeks 4, 16, 24, 48, and 52 of treatment with dupilumab

OTHER OUTCOMES:
Dermatology Life Quality Index (DLQI) | Week 52
  Subject quality of life data will be collected using the DLQI which is a 10-item questionnaire, each question is scored from 0 to 3, giving a total possible score range from 0 to 30, higher score indicating poorer health outcome.
Keloid-Quality of Life Index (K-QLI) questionnaire | Week 52
  Subject quality of life data will be collected using the K-QLI
Keloid distensibility | Week 52
  hardness measured via tonometer
Eczema Area and Severity Index (EASI) score | Week 52
  For those with concomitant atopic dermatitis, disease severity assessments will be performed. The EASI index assigns proportionate values to 4 body regions. Each region is assigned a score of 0 to 3, indicating none, mild, moderate, and severe clinical expression. The percentage of area involved is also assigned an eruption proportional score from 0 to 6. The total body score for each body region is obtained by multiplying the sum of the severity scores by the area score, then multiplying the result by the constant weighted value assigned to that body region. The sum of these scores gives the EASI total from 0-72, with higher score indicating more severity.
Investigator Global Assessment (IGA) of disease score | Week 52
  For those with concomitant atopic dermatitis, disease severity assessments will be performed using the 5 point scale ranging from 0=clear to 4=severe disease
Body Surface Area (BSA) affected with disease | Week 52
  For those with concomitant atopic dermatitis, body surface area affected with AD will be calculated
SCORing Atopic Dermatitis (SCORAD) | Week 52
  For those with concomitant atopic dermatitis, disease severity assessments will be performed. The intensity part of the SCORAD index consists of six items: erythema, edema⁄papulation, excoriations, lichenification, oozing⁄crusts and dryness. Each item graded on a scale 0-3. The subjective items include daily pruritus and sleeplessness, graded on a 10-cm visual analogue scale, with maximum subjective score 20. SCORAD full score is 0-103, with higher score indicating more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT04988022/ICF_001.pdf